CLINICAL TRIAL: NCT03969589
Title: Reproductive Life Planning for Women Veterans With Mental Illness
Brief Title: Reproductive Life Planning for Women With Mental Illness
Acronym: RLP-MH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPO 18-089
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Results first posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Psychotic Disorders; Mood Disorders; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Psychotic Disorders; Mood Disorders; Stress Disorders, Post-Traumatic | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors are blind to participant condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reproductive Life Planning-Mental Health Intervention (Experimental): Reproductive Life Planning-Mental Health (RLP-MH) intervention is comprised of two parts: 1) an in-person interactive session in which the participant works with an RLP-MH facilitator to explore pregnancy intentions and RLP goals, consider important factors that impact those goals (e.g. mental health and physical health conditions, psychosocial and lifestyle factors, values, preferences), and identify personal action steps to address RLP goals and 2) a 15-20 minute follow-up session in person or by phone one month later to discuss progress in addressing RLP goals.
  Interventions: Behavioral: Reproductive Life Planning-Mental Health (RLP-MH) Intervention
- Written materials on Reproductive Life Planning (Other): Participants will receive written materials on reproductive life planning, contraception, and VA resources. Participants will be given the materials and study staff will briefly discuss the content with the participant.
  Interventions: Other: Written Materials on Reproductive Life Planning

INTERVENTIONS:
Behavioral: Reproductive Life Planning-Mental Health (RLP-MH) Intervention — RLP-MH intervention is comprised of two parts: 1) an in-person interactive session in which the participant works with an RLP-MH facilitator to explore pregnancy intentions and RLP goals, consider important factors that impact those goals (e.g. mental health and physical health conditions, psychosocial and lifestyle factors, values, preferences), and identify personal action steps to address RLP goals and 2) a 15-20 minute follow-up session in person or by phone one month later to discuss progress in addressing RLP goals.
  Other Names: RLP-MH
  Arms: Reproductive Life Planning-Mental Health Intervention
Other: Written Materials on Reproductive Life Planning — Participants will receive written materials on reproductive life planning, contraception, and VA resources. Participants will be given the materials and study staff will briefly discuss the content with the participant.
  Arms: Written materials on Reproductive Life Planning

SUMMARY:
Women represent the fastest growing population within the VHA. Many are of reproductive age and experience mental health concerns. Women with mental illness are at greater risk for unplanned pregnancy and poor pregnancy outcomes due to factors related to mental health and mental health treatment. Similarly, mental health concerns (e.g., impact of pregnancy on mental illness, psychiatric medications and pregnancy) can affect reproductive life goals and plans. Reproductive life planning (RLP) interventions that include considerations and concerns women Veterans with mental illness face are needed. The investigators adapted existing RLP materials to create an interactive, individualized, client-centered RLP intervention designed to help women Veterans with mental illness develop a mental health-informed reproductive life plan and reproductive life goals (RLP-MH). The current study aims to determine if the RLP-MH intervention is feasible and acceptable to women Veterans and if it increases engagement in behaviors to address RLP goals.

DETAILED DESCRIPTION:
Many women Veterans are of reproductive age and, of those, a substantial number experience mental health concerns. Women Veterans with mental illness are at greater risk for unplanned pregnancy and adverse pregnancy outcomes due to factors unique to mental illness and mental health treatment. In addition, mental health and mental health-related concerns associated with pregnancy (e.g. impact of pregnancy on mental health, psychiatric medication use during pregnancy) often affect reproductive life decisions and health outcomes. For these reasons, reproductive life planning (RLP), setting personal goals and plans regarding reproductive intentions, that incorporates considerations and addresses concerns specific to mental health conditions is particularly important for women with mental illness. Despite this need, women Veterans with mental illness rarely receive RLP, and current tools do not adequately consider or address the unique reproductive health considerations women with mental illness often experience.

The investigators adapted existing RLP materials to create an interactive, client-centered RLP intervention specifically designed to address mental health considerations that can influence RLP decisions and outcomes in women Veterans with mental illness. Women Veterans work with a facilitator to explore pregnancy intentions and RLP goals; consider important factors that impact those goals (e.g. medical, mental health or psychosocial concerns); and identify steps to address their RLP goals. As such, the RLP-MH intervention may empower women Veterans with mental illness to take an active role in their reproductive health and engage in behaviors that may improve reproductive outcomes. The goal of the proposed study is to pilot-test the RLP-MH intervention in women Veterans with mental illness to evaluate its feasibility and acceptability, and to explore its potential efficacy compared to provision of written materials on RLP (control condition).

ELIGIBILITY:
Inclusion Criteria:

* chart diagnosis of:

  * schizophrenia
  * schizoaffective disorder
  * bipolar disorder
  * major depression
  * PTSD
* current receiving mental health services at one of the recruitment sites

Exclusion Criteria:

* currently pregnant
* inability to have children

  * e.g. infertility, hysterectomy, tubal ligation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Drapalski, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (2):
- United States (2):
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Perry Point VA Medical Center VA Maryland Health Care System, Perry Point, MD, Perry Point, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reproductive Life Planning-Mental Health Intervention | Written Materials on Reproductive Life Planning
Started | 20 | 20
Completed | 17 | 17
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Declined Follow-Up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reproductive Life Planning-Mental Health Intervention | Written Materials on Reproductive Life Planning | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (3.9) | 34.1 (4.7) | 35.0 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 8 | 6 | 14
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Reproductive Life Goal Behavioral Intentions
Description: The Reproductive Life Goal Behavioral Intentions scale was used to measure self-reported intentions to engage in behavior to address one's reproductive life goals. A total score was calculated by taking the sum of the responses to the items. The average total score across participants is reported (range = 1 to 5) with higher scores indicating greater intentions to engage in behaviors to address one's reproductive life goals.
Time Frame: Baseline to 2-Month Post-Intervention (~2 months)
Population: Number analyzed in the rows differ from overall because 3 participants in RLP-MH and 3 in the written materials condition did not complete the 2 month post-treatment assessment
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Reproductive Life Planning-Mental Health Intervention | Written Materials on Reproductive Life Planning
Number analyzed (Participants) | 20 | 20
score on scale
  Baseline | 3.6 (1.3) | 2.7 (1.5)
  2-Month Post Intervention: number analyzed (Participants) | 17 | 17
  2-Month Post Intervention | 3.3 (1.4) | 3.0 (1.7)

2. Primary Outcome: Reproductive Health Decisional Self-Efficacy
Description: The Reproductive Health Decisional Self-Efficacy scale was used to measures expectations or beliefs about one's ability to engage in behaviors that help in making reproductive life decisions. A total score is calculated by taking the sum of response to the items (range = 0 to 44) with higher scores indicating greater decisional self-efficacy.
Time Frame: Baseline to 2-Month Post-Intervention (~2 months)
Population: Number analyzed in the rows differ from overall because 3 participants in RLP-MH and 3 in the written materials condition did not complete the 2-month post-treatment assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reproductive Life Planning-Mental Health Intervention | Written Materials on Reproductive Life Planning
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 35.7 (11.9) | 33.9 (8.8)
  2-Month Post Intervention: number analyzed (Participants) | 17 | 17
  2-Month Post Intervention | 40.7 (3.4) | 38.7 (6.0)

3. Primary Outcome: Attitudes Towards Reproductive Life Planning
Description: The Attitudes Towards Reproductive Life Planning developed for this study will be used to measure attitudes towards reproductive life planning and goal setting across several domains key to effective reproductive life planning. A total score is calculated by taking the sum of responses to the items (range = 7 to 49) with higher scores indicating more positive/favorable attitudes towards reproductive life planning.
Time Frame: Baseline to 2-Month Post-Intervention (~2 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reproductive Life Planning-Mental Health Intervention | Written Materials on Reproductive Life Planning
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 38.1 (12.5) | 42.2 (10.6)
  2-Month Post Intervention: number analyzed (Participants) | 17 | 17
  2-Month Post Intervention | 38.9 (10.8) | 39.4 (11.6)

ADVERSE EVENTS:
Time Frame: Adverse data were collected during their participation in the study (approximately 2 months)
Arm/Group | Reproductive Life Planning-Mental Health Intervention | Written Materials on Reproductive Life Planning
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT03969589/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT03969589/ICF_000.pdf